CLINICAL TRIAL: NCT04965636
Title: A Phase 3, 52-week, Open-label, Single Arm Study to Investigate the Efficacy and Safety of Mepolizumab SC in Participants Aged 6 to 17 Years With Hypereosinophilic Syndrome
Brief Title: Study in Pediatrics With HypEREosinophilic Syndrome (SPHERE)
Acronym: SPHERE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215360
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Hypereosinophilic Syndrome; Mepolizumab; Safety; Efficacy; Pediatric; Adolescent
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: This is a single arm study
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving mepolizumab (Experimental)
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab will be provided in pre-filled safety syringe

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of mepolizumab in children and adolescents with hypereosinophilic syndrome (HES) who are receiving standard of care (SoC) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be aged 6 to 17 years inclusive, at Screening (Visit 1).
* Participants who have been diagnosed with HES for at least 6 months prior to enrolment (Visit 2).
* A history of 2 or more HES flares within the past 12 months prior to Screening (Visit 1).
* Participants must have blood eosinophil count >=1000 cells per microliter (/mcL) present at Screening.
* Participants must be on a stable dose of HES therapy for the 4 weeks prior to the first dose of mepolizumab (Visit 2)
* Male and/or female
* Signed written informed consent

Exclusion Criteria:

* Life-threatening HES or life-threatening HES co-morbidities
* Other concurrent medical conditions that may affect the participant's safety
* Eosinophilia of unknown significance
* Fusion tyrosine kinase gene translocation [FIP1L1- Platelet-derived Growth Factor Receptor (PDGFRα) (F/P)] positivity
* Clinical diagnosis of eosinophilic granulomatosis with polyangiitis (EGPA)
* Participants with chronic or ongoing active infections requiring systemic treatment, as well as participants who have experienced clinically significant infections due to viruses, bacteria, and fungi within 4 weeks prior to enrolment (Visit 2)
* Participants with a pre-existing parasitic infestation within 6 months prior to enrolment (Visit 2)
* Participants with a known immunodeficiency (e.g. Human immunodeficiency virus [HIV]), other than that explained by the use of OCS or other therapy taken for HES
* Participants with documented history of any clinically significant cardiac damage prior to Screening (Visit 1) that, in the opinion of the investigator, would impact the participant's participation during the study
* Participants with a history of or current lymphoma, Participants with current malignancy or previous history of cancer in remission for less than 12 months prior to Screening (Visit 1)
* Participants who are not responsive to OCS based on clinical response or blood eosinophil counts.
* Participants who have previously received mepolizumab in the 4 months prior to enrolment (Visit 2)
* Participants receiving non-oral systemic corticosteroids in the 4-week period prior to enrolment (Visit 2).
* Participants who have received any other monoclonal antibodies within 30 days or 5 half-lives, whichever is longer, of enrolment (Visit 2).
* Participants who have received treatment with an investigational agent (biologic or non-biologic) within the past 30 days or 5 drug half-lives, whichever is longer, prior to enrolment (Visit 2).
* Use of candidate Coronavirus disease 2019 (COVID-19) vaccines that have not received limited, accelerated, or full authorization/approval, and are only in use as part of a clinical trial.
* Participants who are currently participating in any other interventional clinical study
* Participants with any history of hypersensitivity to any monoclonal antibody (including mepolizumab).
* Evidence of clinically significant abnormality in the hematological, biochemical, or urinalysis screen from the sample collected at Screening (Visit 1), that could put the participant's safety at risk by participating in the study, as judged by the investigator

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Number of HES flares experienced by participants per year | Up to Week 52
  The annualized rate of HES flares will be measured.

SECONDARY OUTCOMES:
Change in mean daily oral corticosteroids (OCS) dose (prednisone/prednisolone or equivalent) from Weeks 0 to 4 to Weeks 48 to 52 | Weeks 0 to 4 and Weeks 48 to 52
  Change in mean daily OCS dose (prednisone/prednisolone or equivalent) will be assessed.
Number of participants with >=50 percent (%) reduction in mean daily OCS dose (prednisone/prednisolone or equivalent) from Weeks 0 to 4 compared with Weeks 48 to 52 | Weeks 0 to 4 and Weeks 48 to 52
  Number of participants with >=50% reduction in mean daily OCS dose (prednisone/prednisolone or equivalent) will be assessed.
Number of participants achieving a mean daily OCS dose (prednisone/prednisolone or equivalent) of <=7.5 milligrams (mg) during Weeks 48 to 52 in participants that are taking OCS at Baseline | Weeks 48 to 52
  Number of participants achieving a mean daily OCS dose (prednisone/prednisolone or equivalent) of <=7.5 mg will be assessed.
Number of participants achieving a mean daily OCS dose (prednisone/prednisolone or equivalent) of <=7.5 mg during Weeks 48 to 52 | Weeks 48 to 52
  Participants achieving mean daily OCS dose (prednisone/prednisolone or equivalent) of <=7.5 mg will be evaluated.
Change from Baseline in fatigue severity based on Brief Fatigue Inventory (BFI) Item 3 (worst level of fatigue during past 24 hours) for Week 52 | Baseline and up to Week 52
  Item 3 of the BFI is a 11-point scale that measures fatigue (weariness, tiredness) ranging from 0 "no fatigue" to 10 "as bad as you can imagine".
Number of participants with Anti-drug antibodies (ADA) and neutralizing antibodies (NAb) | Up to Week 52
  Participants with ADA and NAb will be evaluated.
Ratio to Baseline in absolute blood eosinophil count | Baseline and up to Week 52
  Blood samples will be collected.
Mepolizumab plasma concentrations | Week 4 and up to Week 52
  Blood samples will be collected for determination of mepolizumab plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (4):
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Charleston, South Carolina
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Quilmes
- Brazil (2):
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Sorocaba
- GSK Investigational Site, Petah Tikva, Israel
- GSK Investigational Site, Rotterdam, Netherlands
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com